CLINICAL TRIAL: NCT05230290
Title: Evaluation of Safety, Tolerability, and Pharmacokinetics of KD6001 in Patients With Advanced Solid Tumours - Phase I Clinical Study
Brief Title: Clinical Study of KD6001 in Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Kanda Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD6001CT01
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD6001 Injection (Experimental): Participants will be administered KD6001 at an applicable dose as monotherapy
  Interventions: Biological: KD6001 Injection

INTERVENTIONS:
Biological: KD6001 Injection — Solution for intravenous injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and clinical activity of KD6001 as treatment for participants with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Being voluntary to sign the informed consent form.
* Age ≥ 18 and ≤ 70 years at the time of signing informed consent form, male or female.
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
* Patients with histologically or cytologically confirmed advanced solid tumors: patients with advanced solid tumors who have failure in standard of care, cannot tolerate standard of care, refuse and/or have no standard of care (melanoma, renal carcinoma and urothelial carcinoma).
* Patients with at least one measurable lesion at baseline according to RECIST (Version 1.1).
* Agree to provide tumor tissue specimen (fresh biopsied sample before treatment should be provided as far as possible, the archived sample within two years is acceptable for the patients who cannot provide fresh biopsied sample before treatment).
* Adequate organ function as indicated by the laboratory results during the screening period.
* Use of highly-effective contraceptive methods during the whole study for men of reproduction ability or women of pregnant possibility (e.g. oral contraceptives, intrauterine contraceptive device or barrier contraception in combination with spermatocide), and continuation of contraception for 6 months after the end of study treatment.
* Good compliance, cooperation with follow-up.

Exclusion Criteria:

* Subjects with history of other malignant tumors within the five years prior to study entry. Except for the malignant tumors that can be expected to be cured after treatment (including treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated by radical surgery).
* Have been previously exposed to any anti-tumor treatment, or local anti-tumor treatment, or received investigational drug or instrument therapy.
* Having received immunotherapy within 8 weeks prior to first dose of study drug (including antibody therapy and cell therapy); Subjects with prior anti-CTLA-4 checkpoint inhibitors should be excluded.
* Adverse reaction induced by previous therapy having not recovered to CTCAE (version 5.0) grade 1 or better (except alopecia and neurotoxicity, which is determined by investigators that long-term presence could not be restored).
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Having central nervous system metastases and/or cancerous meningitis.
* Subjects with previously treated brain metastases may participate.
* Having or suspected to have active autoimmune disease.
* Patients with severe hepatitis and liver cirrhosis.
* Massive hydrothorax or ascites with clinical symptoms or requiring symptomatic treatment; Having serious cardiovascular diseases, pulmonary diseases, interstitial pneumonia, chronic obstructive pulmonary disease, and symptomatic bronchospasm heart disease; Having active infection requiring systemic treatment; Positive test for HIV or AIDS; chronic active HBV or HCV; Patients with active tuberculosis.
* Systemic glucocorticoids (prednisone > 10 mg / day or other glucocorticoids of equivalent dose) and other immuno-suppressive drugs were used within 14 days before the first study drug treatment; Use of broad-spectrum antibiotics that may affect the change of intestinal flora within 14 days prior to the first dose of study drug.
* Vaccination of live vaccine within 4 weeks prior to the start of study; Having received major surgery within 4 weeks prior to the first dose of study drug; History of anti-psychotics abuse and unable to abstain, or with a history of mental disorder.
* Pregnant or breastfeeding women.
* Allergy to KD6001 or its excipients.
* Other severe, acute or chronic medical diseases or abnormalities in laboratory examination possibly increasing the relevant risk in study participation or possibly interfering the interpretation of study results as judged by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to Day 28
  DLTs will be assessed during the dose-escalation phase and are defined as toxicities.
Incidence and nature of participants with adverse events (AEs) | Baseline until 30 days after last dose of KD6001
  Evaluate the adverse events (AE) according to NCI CTCAE 5.0.
To determine the Maximum tolerated dose (MTD)/Recommended Phase II dose (RP2D) of KD6001 in subjects with solid tumors | Baseline to study completion up to 2 years
  If more than or equal to one third of the participants at a dose level experience dose limiting toxicity (DLT), the MTD reassessed and the next lowest dose level for the combination therapy considered the MTD.

SECONDARY OUTCOMES:
Antitumor activity measured by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST)/Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Baseline to study completion up to 2 years
  Number of participants with response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Descriptive statistics and graphical analysis will be used to summarize patients' demographic and clinicopathological characteristics, patient safety and efficacy outcomes and correlative markers.
To characterize the pharmacokinetics (PK) profile of KD6001: Maximum Observed Concentration (Cmax) | Baseline to study completion up to 2 years
  Serum concentrations of KD6001 in individual subjects at different time points after KD6001 administration
To evaluate the immunogenicity of KD6001: Number of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline until 15 days after last dose of KD6001
  The immunogenicity of KD6001 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China